CLINICAL TRIAL: NCT00939666
Title: Minimal Invasive Treatment for Patients With Good Response to Chemoradiation With Selection and Follow-up by MRI: a Single Arm Phase-II Feasibility Study in Rectal Cancer
Brief Title: Minimal Invasive Strategies for Good and Complete Response to Chemoradiation in Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC 09-2-034
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Rectal cancer; Chemoradiation; Response; Wait-and-see policy; Transanal endoscopic microsurgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wait&see or TEM with intensive follow-up (Experimental): All patients will be included in this arm
  Interventions: Procedure: Wait&see or TEM with intensive follow-up

INTERVENTIONS:
Procedure: Wait&see or TEM with intensive follow-up — Wait&see or TEM with intensive follow-up

SUMMARY:
The high proportion of complete and good responders with modern chemoradiation and the improvement in magnetic resonance (MR)-imaging techniques have stimulated a renewed interest to the question whether in patients with complete or good response the overall benefits of a 'wait-and-see policy' or transanal endoscopic microsurgery (TEM) combined with intensive follow-up may outweigh the benefits associated with conventional surgery (total mesorectal excision (TME)or abdominoperineal resection (APR)). On the one hand, less invasive strategies will expose subjects to more diagnostic procedures and possibly a slightly higher risk of local failure and the need for salvage surgery. On the other hand, mortality and morbidity associated with radical surgery (e.g. anastomotic leakage, relaparotomy, wound and pelvic infection, chronic wound healing disturbances, abscess, colostomy, faecal or urinary incontinence and sexual dysfunction) can be avoided. The investigators believe that wait-and-see policy for complete responders and TEM for good responders after chemoradiation is a feasible alternative to standard surgery, provided these patients are intensively followed.

DETAILED DESCRIPTION:
The high proportion of complete and good responders with modern chemoradiation and the improvement in magnetic resonance (MR)-imaging techniques have stimulated a renewed interest to the question whether in patients with complete or good response the overall benefits of a 'wait-and-see policy' or transanal endoscopic microsurgery (TEM) combined with intensive follow-up may outweigh the benefits associated with conventional surgery (total mesorectal excision (TME) or abdominoperineal resection (APR)). On the one hand, less invasive strategies will expose subjects to more diagnostic procedures and possibly a slightly higher risk of local failure and the need for salvage surgery. On the other hand, mortality and morbidity associated with radical surgery (e.g. anastomotic leakage, relaparotomy, wound and pelvic infection, chronic wound healing disturbances, abscess, colostomy, faecal or urinary incontinence and sexual dysfunction) can be avoided. The investigators believe that wait-and-see policy for complete responders and TEM for good responders after chemoradiation is a feasible alternative to standard surgery, provided these patients are intensively followed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients with primary rectal cancer without distant metastases who underwent CRT and show clinical complete response or very good response: Clinical complete response (ycT0N0) or very good response (ycT1-2N0) after pre-operative chemoradiation will be determined clinically (digital rectal examination, endoscopy), radiologically (contrast-enhanced-MRI) and pathologically (biopsy)
* Informed consent and capability of giving informed consent
* Comprehension of the alternative strategies and the concept of unknown risks are clear to the patient (in other words that the patient understands the experimental base of the study).

Exclusion Criteria:

* Recurrent rectal cancer.
* Distant metastasis.
* Unable or unwilling to comply to the intensive follow-up schedule.
* Contra-indications for MRI. If MRI is not possible because of contra-indications (e.g. pacemaker) we will exclude patients. MRI is crucial for response evaluation and follow-up and can not be omitted in patients that follow the alternative strategies ('wait-and-see policy' or TEM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07-01; Primary Completion 2014-09-01 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Local recurrence | 2 and 5 years

SECONDARY OUTCOMES:
Overall survival | 2 and 5 years
Disease-free survival | 2 and 5 years
Distant metastasis-free survival | 2 and 5 years
Quality of life | 6 weeks to 1 year
Compliance | 2 and 5 years
Percentage of patients that chooses the minimal invasive strategies over standard surgery | 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Geerard L Beets, MD, PhD, Principal Investigator — Maastricht University Medical Center, Maastricht, The Netherlands
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Laurentius Hospital Roermond, Roermond

IPD SHARING:
Plan to Share IPD: Undecided
Pooling of data is expected in the future

REFERENCES:
- [Result] Maas M, Beets-Tan RG, Lambregts DM, Lammering G, Nelemans PJ, Engelen SM, van Dam RM, Jansen RL, Sosef M, Leijtens JW, Hulsewe KW, Buijsen J, Beets GL. Wait-and-see policy for clinical complete responders after chemoradiation for rectal cancer. J Clin Oncol. 2011 Dec 10;29(35):4633-40. doi: 10.1200/JCO.2011.37.7176. Epub 2011 Nov 7. PMID 22067400
- [Derived] Haak HE, Zmuc J, Lambregts DMJ, Beets-Tan RGH, Melenhorst J, Beets GL, Maas M; Dutch Watch-and-Wait Consortium. The evaluation of follow-up strategies of watch-and-wait patients with a complete response after neoadjuvant therapy in rectal cancer. Colorectal Dis. 2021 Jul;23(7):1785-1792. doi: 10.1111/codi.15636. Epub 2021 Apr 2. PMID 33725387